CLINICAL TRIAL: NCT05005663
Title: Incisional Hernia in Children and and Infants : a Tertiary Center Experience
Brief Title: Incisional Hernia in Infants and Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammad Gharieb Mohammad Khirallah, assistant professor of pediatric surgery, Tanta University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 34687/5/21
Record Dates: First submitted 2021-08-05; First posted 2021-08-13 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Incisional Hernia
Keywords: incisional hernia; infants; children; tissue repair; wound healing
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): patients younger than 2 years
  Interventions: Other: surgical management of incisional hernia
- group B (Active Comparator): patients older than 2 years
  Interventions: Other: surgical management of incisional hernia

INTERVENTIONS:
Other: surgical management of incisional hernia — surgical repair of the incisional hernia

SUMMARY:
the study of development of incisional hernia in infants and children at a tertiary level experience.

DETAILED DESCRIPTION:
Background: incisional hernia in children and infants (IHCI) represents a major complication following exploration. The condition is associated with prolonged hospital stay, readmission and the need for another operation to treat the resulting incisional hernia. The incidence is variable worldwide. The leading causes are still indeterminate as well as the management strategy. We aimed at studying IHCI at a tertiary level hospital as regard presenting symptoms, methods of management and its impact on the quality of life of patients.

Methods: a retrospective study included all infants and children presented with incisional hernia. Patients were categorized in to two groups according to the age of presentation, group A patients younger than two years of age and group B patients older than two years. All data related to the first operation in addition to data related to repair of the incisional hernia were collected in special charts.

ELIGIBILITY:
Inclusion Criteria:

* all infants and children with incisional hernia

Exclusion Criteria:

* congenital abdominal wall defects

Ages: 8 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 67 (Estimated)
Dates: Start 2007-02-02 (Actual); Primary Completion 2022-12-20 (Estimated); Study Completion 2023-01-22 (Estimated)

PRIMARY OUTCOMES:
repair of incisional hernia | 2 years
  surgical repair

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Tanta, Egypt